CLINICAL TRIAL: NCT02150993
Title: A Randomized, Non-comparative, Phase IIb, Unblinded Trial, Evaluating the Efficacy and Safety of Tenofovir-emtricitabine or Lamivudine Plus Zidovudine, Lopinavir/Ritonavir, or Raltegravir, Among ARV-naïve HIV-2 Infected Adult Patients, in West Africa
Brief Title: First-Line Treatment for HIV-2
Acronym: FIT-2
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 12294 FIT-2
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: HIV-2 Infection
Keywords: Africa; Antiretroviral Treatment; HIV-2; firsts line ART; Adults
MeSH Terms: interventions — Tenofovir; Emtricitabine; Lamivudine; Zidovudine; Lopinavir; Ritonavir; Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A : TDF + FTC (or 3TC) + ZDV (Experimental): Tenofovir + Emtricitabine or Lamivudine + Zidovudine
  Interventions: Drug: Tenofovir + Emtricitabine or Lamivudine + Zidovudine
- TDF+FTC (or 3TC) +LPV/r (Experimental): Tenofovir + Emtricitabine or Lamivudine + Lopinavir/ritonavir
  Interventions: Drug: Tenofovir + Emtricitabine or Lamivudine + Lopinavir/ritonavir
- Arm C : TDF +FTC (or 3TC) + RAL (Experimental): Tenofovir + Emtricitabine or Lamivudine + Raltegravir
  Interventions: Drug: Tenofovir + Emtricitabine or Lamivudine + Raltegravir

INTERVENTIONS:
Drug: Tenofovir + Emtricitabine or Lamivudine + Zidovudine — TDF +FTC or 3TC (Tenofovir disoproxil fumarate 245 mg and emtricitabine 200 mg or lamivudine 300mg) QD (evenings orally with meals) + ZDV (Zidovudine 300 mg) 1 tb BID (mornings and evenings orally)
  Other Names: TDF+FTC (or 3TC) + ZDV; TDF+FTC (or 3TC) + AZT
  Arms: Arm A : TDF + FTC (or 3TC) + ZDV
Drug: Tenofovir + Emtricitabine or Lamivudine + Lopinavir/ritonavir — TDF +FTC or 3TC (Tenofovir disoproxil fumarate 245 mg and emtricitabine 200 mg or lamivudine 300mg) QD (evenings orally with meals) + Lop/r (Lopinavir/ritonavir lopinavir 200/50 mg) 2 tbs BID (mornings and evenings orally)
  Other Names: TDF +FTC (or 3TC) +LPV/r
  Arms: TDF+FTC (or 3TC) +LPV/r
Drug: Tenofovir + Emtricitabine or Lamivudine + Raltegravir — TDF +FTC or 3TC (Tenofovir disoproxil fumarate 245 mg and emtricitabine 200 mg or lamivudine 300mg) QD (evenings orally with meals) + RAL (Raltegravir 400 mg) 1 tb BID (mornings and evenings orally)
  Other Names: TDF +FTC (or 3TC) + RAL
  Arms: Arm C : TDF +FTC (or 3TC) + RAL

SUMMARY:
FIT-2 is a multi-country, phase IIb, randomized, non-comparative study, carried out in West Africa (Côte d'Ivoire, Burkina Faso, Senegal, Togo).

ARV-naïve HIV-2 infected adult patients will be recruited and followed during 96 weeks.

The objective is to evaluate the efficacy and safety of 3 first-line treatments in HIV-2 infected adult patients, in West Africa. A treatment will be considered as effective if more than 55% of patients in that arm attain "global success" at 96 weeks.

DETAILED DESCRIPTION:
Main objective

To determine in treatment-naïve HIV-2 infected patients, with CD4 counts above 200 cells/mm3, which of the following three regimens of first line treatment, Tenofovir (TDF), Emtricitabine or lamivudine (FTC or 3TC) plus Zidovudine (ZDV); TDF-FTC (3TC) plus Lopinavir/ritonavir (LPV / r); or TDF-FTC (3TC) plus raltegravir (RAL), will result in an "global success" rate of > 55% at week 96.

Number of participants : 210

Main outcome :

The proportion of patients with "global success" at W96, defined by survival with a plasma HIV-2 RNA viral load of <50 copies/ml and the non-occurrence of AIDS classified events (excluding tuberculosis) and the non-occurrence of severe morbidities non-AIDS-defining illness (cardiovascular disease, kidney disease, severe bacterial disease) and a delta of CD4 depending on the initial CD4 count (CD4 delta > +100cells/mm3 for initial CD4s between 201 and 500 cells/mm3 or delta ≥0 cells/mm3 for initial CD4s > +500 cells/mm3)

Inclusion criteria:

* Infection by HIV-2 only;
* Age > or = 18 years;
* Naïve for antiretroviral therapy (including antiretroviral treatment in the context of PMTCT except taking a dose of Nevirapine for PMTCT)
* CD4 >200 cells/mm3
* Resident of the city where the study is held or of city suburbs to facilitate participation
* Signed informed consent document

ELIGIBILITY:
Inclusion Criteria:

* Infection by HIV-2 only;
* Age > ou = 18 years;
* Naïve for antiretroviral therapy (including antiretroviral treatment in the context of PMTCT except taking a dose of Nevirapine for PMTCT)
* CD4 >200 cells/mm3
* Resident of the city where the study is held or of city suburbs to facilitate participation
* Signed informed consent document

Exclusion Criteria:

* Current participation in any other clinical trial
* Presence of opportunistic non-stabilized infections, of any serious or progressive disease, or of any clinical signs consistent with severe disease whose diagnosis is not yet confirmed, such as fever, weight loss, diarrhea or cough not yet explained (non-exhaustive list).
* All pathology that leads in daily life to prefer one or the other of the three therapeutic regimens for medical reasons or to change the dosages specified in the test. This includes (but not limited to):
* Hemoglobin ≤ 8 g / dL
* Neutrophil count <500 cells/mm3
* Renal impairment with creatinine clearance <50mL/mn
* Blood platelet <50 000 cells/mm3
* Decompensated heart failure
* Hepatic failure Severe (TP<50% or cytolysis severe (ALAT> 3x ULN)
* Active TB during treatment with rifampicin
* Taking drugs that interact with the drugs of the clinical trial (as specified in the SPC)
* Pregnancy, breastfeeding or planning to become pregnant during study follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2016-01-26 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
The "overall success" | 96 weeks
  The proportion of patients with "global success" at W96, defined by survival with a plasma HIV-2 RNA viral load of <50 copies/ml and the non-occurrence of AIDS classified events (excluding tuberculosis) and the non-occurrence of severe morbidities non-AIDS-defining illness (cardiovascular disease, kidney disease, severe bacterial disease) and a delta of CD4 depending on the initial CD4 count (CD4 delta> +100cells/mm3 for initial CD4s between 201 and 500 cells/mm3 or delta ≥0 cells/mm3 for initial CD4s > +500 cells/mm3)
  A treatment is considered to be effective if the "global success" is > 55 % at 96 weeks.

SECONDARY OUTCOMES:
Therapeutic failure | 24 weeks
  The percentage of patients in "treatment failure" defined by :
  1. death or
  2. a delta ≤0 CD4 cells / mm3 between W2 and W24 (or W48) for patients with baseline CD4 between 201 and 500 cells / mm3 or if % of decrease in CD4 > 20% between W2 and W24 (or W48) for patients with baseline CD4 > 500 cellules/mm3 or
  3. a plasma HIV-2 RNA viral load of > or =50 copies/ml or
  4. the occurrence of an AIDS defining event (excluding tuberculosis).
Therapeutic failure | 48 weeks
  The percentage of patients in "treatment failure" defined by :
  1. death or
  2. a delta ≤0 CD4 cells / mm3 between W2 and W24 (or W48) for patients with baseline CD4 between 201 and 500 cells / mm3 or if % of decrease in CD4 > 20% between W0 and W24 (or W48) for patients with baseline CD4 > 500 cellules/mm3 or
  3. a plasma HIV-2 RNA viral load of > or = 50 copies/ml or
  4. the occurrence of an AIDS defining event (excluding tuberculosis).
Incidence and type of severe clinical or biological severe adverse events per arm | between Week 0 and Week 96
  Incidence and type of severe clinical or biological severe adverse event (grade 3 or 4)
The clinical progression | between Week 0 and Week 96
  The incidence of severe morbidity, defined as: AIDS morbidity, non-AIDS cancer, severe non-AIDS bacterial disease, or any disease leading to death
The evolution of CD4 counts | between Week 0 and Week 96
  Evolution of the absolute and percentage CD4 counts during follow-up
The evolution of plasma HIV-2 RNA load | between at W0 and W96
  Evolution of the plasma viral load during follow-up
The observance of antiretroviral treatment | between W0 and W96
  To describe the antiretroviral possession ratio and assessment of compliance by questionnaire
The resistance mutations profile | Weeks 96
  Description of new resistance mutations profiles in cases of treatment failure
The evolution of the HIV-2 DNA titers in PBMC | between Week 0 and Week 96
  To describe the evolution the HIV-2 DNA titers in PBMC
The frequency of treatment switches and discontinuations | between Week 0 and Week 96
  The frequency of modifications and discontinuations of treatment per arm
To model the long-term survival and cost-effectiveness ratio | Weeks 96
  The probability of survival and the incremental cost-effectiveness of these three treatment regimens

CONTACTS AND LOCATIONS:
Overall Officials: Serge P. Eholié, MD, MSc, Pr, Principal Investigator — Service des Maladies Infectieuses et Tropicales, CHU de Treichville, Abidjan, Côte d'Ivoire; Françoise P. Brun-Vézinet, MD, MSc, Pr, Principal Investigator — Laboratoire de virologie, Hôpital Bichat-Claude Bernard
Locations (9):
- Burkina Faso (2):
  - CHU Sourô Sanou, Bobo-Dioulasso
  - CHU Yalgado Ouedraogo, Ouagadougou
- Côte d’Ivoire (5):
  - Centre de Prise en Charge et de Formation (CePReF), Association ACONDA, Abidjan
  - Centre Médical du Suivi des Donneurs de Sang (Blood Bank Medical Centre), Abidjan
  - CIRBA, Abidjan
  - o L'Unité de soins ambulatoires et de conseils (USAC), CHU de Treichville, Abidjan
  - Service des Maladies Infectieuses et Tropicales (SMIT), CHU de treichville, Abidjan
- CHNU Fann, Dakar, Senegal
- ONG Espoirs Vie Togo (EVT), Lomé, Togo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Eholie SP, Ekouevi DK, Chazallon C, Charpentier C, Messou E, Diallo Z, Zoungrana J, Minga A, Ngom Gueye NF, Hawerlander D, Dembele F, Colin G, Tchounga B, Karcher S, Le Carrou J, Tchabert-Guie A, Toni TD, Ouedraogo AS, Bado G, Toure Kane C, Seydi M, Poda A, Mensah E, Diallo I, Drabo YJ, Anglaret X, Brun-Vezinet F; FIT-2 study group. Efficacy and safety of three antiretroviral therapy regimens for treatment-naive African adults living with HIV-2 (FIT-2): a pilot, phase 2, non-comparative, open-label, randomised controlled trial. Lancet HIV. 2024 Jun;11(6):e380-e388. doi: 10.1016/S2352-3018(24)00085-7. Epub 2024 May 10. PMID 38740027
- See also: sponsor site — http://www.anrs.fr
- See also: Related Info — http://www.mereva.net/